CLINICAL TRIAL: NCT04523350
Title: Randomized Multi-Center, Subject and Evaluator Blinded, Parallel-Group Study to Evaluate the Safety and Effectiveness of the Instylla Hydrogel Embolic System (HES) Compared With Standard of Care Transcatheter Arterial Embolization (TAE) / Transcatheter Arterial Chemoembolization (cTACE) for Vascular Occlusion of Hypervascular Tumors; A Pivotal Study
Brief Title: Instylla HES Hypervascular Tumor Pivotal Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instylla, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: INY-P-20-001
Record Dates: First submitted 2020-08-17; First posted 2020-08-21 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-12

CONDITIONS: Hypervascular Tumors

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Instylla HES (Experimental)
  Interventions: Device: Instylla HES
- Control (Active Comparator): TAE or cTACE
  Interventions: Other: TAE or cTACE

INTERVENTIONS:
Device: Instylla HES — Instylla HES is a novel liquid embolic made of primarily water and polyethylene glycol (PEG)
  Arms: Instylla HES
Other: TAE or cTACE — Bland TAE or cTACE
  Other Names: Control
  Arms: Control

SUMMARY:
To determine whether Instylla HES has the ability to effectively embolize targeted arterial segments of hypervascular tumors as well as (i.e., is non-inferior to) standard of care (SOC) transarterial embolization/conventional transarterial chemoembolization, while resulting in an acceptable risk of device and procedure-related serious adverse events.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects age ≥ 22 years old
2. Subjects with confirmed finding of hypervascular tumor on CT and/or MRI for whom TAE or cTACE is medically indicated, including but not limited to:

   1. Subjects with unresectable primary or metastatic hepatic cancer
   2. Subjects with primary, metastatic or benign renal tumors
   3. Subjects with bone metastases
   4. Subjects with adrenal tumors
   5. Subjects with other hypervascular tumors
3. Subjects with at least one target lesion that is well-delineated such that, in the Investigator's opinion, the lesion can be measured in at least one dimension as 1 cm or more, suitable for remeasurement, and demonstrating definitive arterial enhancement (Note: Pre-operative tumors do not need to meet this criterion.)
4. Subjects with at least one target vessel ≤ 5mm and Instylla HES can be delivered to the target vessel(s).
5. Eastern Cooperative Oncology Group Performance Status (ECOG PS) of 0-2 (PS 0-1 for metastatic disease)
6. Subject or authorized representative have been informed of the nature of the study and has provided written informed consent approved by the appropriate local Ethics Committee/Institutional Review Board and agrees to comply with all protocol specified follow-up appointments.
7. Expected life expectancy ≥ 6 months after Index embolization

Exclusion Criteria:

1. Embolization for lesions other than hypervascular tumors such as arteriovenous malformations.
2. It is anticipated that not all target vessels requiring embolization during the index procedure can be embolized with either HES alone or the SOC embolization agent as assigned.
3. Undergoing radioembolization or DEB-TACE for Index Procedure
4. Undergoing a planned secondary procedure the same day as the Index Procedure
5. Requires TAE/cTACE for liver tumors via extrahepatic collateral artery(ies)
6. Prior radioembolization of the target tumor lesion/vascular bed within 30 days of the Index Procedure.
7. For subjects with HCC or undergoing embolization to the liver: Child-Pugh Class C or presence of complete portal vein thrombosis.
8. Tumor lesions > 8 cm in diameter (in one direction) or >50% tumor volume burden of the target organ
9. If subject was treated with Avastin, last dose is within 4 weeks of the planned procedure.
10. Known severe atheromatosis or vascular anatomy that precludes catheterization
11. Presence of bilioenteric anastomoses and/or prior biliary stenting/drainage or any violation of the biliary sphincter, including sphincterotomy for embolization of liver tumors
12. Target lesion supplied by the pulmonary artery, coronary artery, or cerebral or cerebellar artery (requiring embolization of these arteries) or the artery to be embolized has connections to these arteries via a collateral pathway
13. Known allergies (based on history) to PEG, ferrous compounds, tert Butyl Hydroperoxide, contrast media or procedural sedatives/anesthetics that is not amenable to pre-medication
14. Uncorrectable impaired clotting: Platelet count <30,000/µL or International Normalized Ratio (INR) > 1.5
15. Serum creatinine > 2 mg/dL
16. Serum bilirubin level > 3 mg/dL
17. Serum albumin < 2.5 g/dL
18. Any contraindication to angiography or embolization protocol utilized at treating institution.
19. Pregnant or breast-feeding or females planning on becoming pregnant with the next 3 months (women of child-bearing potential must undergo a pregnancy test performed in accordance with local institutional requirements).
20. Other concurrent conditions including an ongoing adverse effect or complication of prior therapy or adverse drug reactions, that in the opinion of the Investigator or Clinical Events Committee, would be unlikely to receive clinical benefit from the study procedure or participation in the study may compromise subject safety or study objectives (including but not limited to ongoing acute infection, renal dysfunction, morbid obesity, severe cardiac disease).
21. Enrollment in a concurrent study in which the study treatment may confound the evaluation of the study device

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2021-01-04 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2024-11-19 (Actual)

PRIMARY OUTCOMES:
Primary Effectiveness Endpoint: Delivery of the embolic agent to the index tumor feeding vessel with stasis of flow as determined by an independent radiologist via comparison of the pre and final post procedure images | Immediately post-embolization procedure
  Stasis of flow defined as absence of contrast flow within the targeted tumor feeding vessel
Primary Safety Endpoint: Freedom from major adverse events through 30 days post-index procedure | 30 days post-embolization procedure

CONTACTS AND LOCATIONS:
Overall Officials: Nadine Abi-Jaoudeh, M.D., Principal Investigator — University of California, Irvine
Locations (15):
- United States (12):
  - UAB Hospital, Birmingham, Alabama
  - Central Arkansas Radiation Therapy Institute, Inc., Little Rock, Arkansas
  - University of California, Irvine, Irvine, California
  - Memorial Health Services, Long Beach, California
  - Olive View-UCLA Education & Research Institute, Sylmar, California
  - St. Elizabeth Healthcare, Edgewood, Kentucky
  - Boston Medical Center, Boston, Massachusetts
  - Summit Health, Florham Park, New Jersey
  - New York and Presbyterian Hospital (Cornell/Weill Medical College), New York, New York
  - Charlotte Radiology, Charlotte, North Carolina
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania
- Canada (3):
  - Sunnybrook Research Institute, Toronto, Ontario
  - Mount Sinai, Toronto, Ontario
  - Toronto General Hospital, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No